CLINICAL TRIAL: NCT01339273
Title: Ultrasound Guided Transversus Abdominis Plane (TAP) Block for Postoperative Analgesia After Laparoscopic Colonic Resection- a Double Blind Randomised Controlled Trial
Brief Title: Transversus Abdominis Plane (TAP) Block for Postoperative Analgesia After Laparoscopic Colonic Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Nicholas Crabtree, Consultant Anaesthetist, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sponsorship review number:113
Record Dates: First submitted 2011-04-18; First posted 2011-04-20 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Colonic Cancer; Rectal Cancer; Colonic Diverticulum; Ulcerative Colitis
Keywords: TAP block; Laparoscopic hemicolectomy; Laparoscopic anterior resection; laparoscopic colonic resection
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Diverticulum, Colon; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP block (Experimental): Patients in this arm will receive ultrasound guided TAP bock with Bupivacaine 0.25% 20ml per side or to a maximum 1mg/kg per side and the skin puncture will be covered with a small plaster
  Interventions: Procedure: Ultrasound guided Transversus Abdominis Plane (TAP) bock
- Local anaesthetic infiltration (Active Comparator): Laparoscopic port sites and specimen extraction site will be infiltrated with a total of 40 mls 0.25% bupivacaine subcutaneously at the end of the procedure in the control group and plasters will be stuck on either side approximately where a skin puncture for tap block would be made.
  Interventions: Procedure: Local anaesthetic infiltration of laparoscopic port sites

INTERVENTIONS:
Procedure: Ultrasound guided Transversus Abdominis Plane (TAP) bock — Ultrasound guided TAP bock with Bupivacaine 0.25% 20ml per side or to a maximum 1mg/kg per side and the skin puncture will be covered with a small plaster
  Arms: TAP block
Procedure: Local anaesthetic infiltration of laparoscopic port sites — Laparoscopic port sites and specimen extraction site will be infiltrated with a total of 40 mls 0.25% bupivacaine subcutaneously at the end of the procedure in the control group and plasters will be stuck on either side approximately where a skin puncture for tap block would be made.
  Arms: Local anaesthetic infiltration

SUMMARY:
Laparoscopic (key-hole) large bowel resection is a minimally invasive procedure when compared to open large bowel resection, but is still associated with a significant amount of pain and discomfort. Analgesia is commonly provided by a multi-modal technique involving varying combinations of paracetamol, Non steroidal anti-inflammatory drugs (NSAIDs), regional analgesia and oral or parenteral opioids. While epidural analgesia is considered the gold standard for open colo-rectal procedures it can be associated with significant complications and may delay hospital discharge in laparoscopic procedures. Opioids are associated with an increased incidence of nausea, vomiting and sedation and reduced bowel motility which can also prolong recovery.

Transversus Abdominis Plane (TAP) block is a technique which numbs the nerves carrying pain sensation from the abdominal wall and provides effective and safe analgesia with minimal systemic side effects. Their perceived benefits are thought to relate to reduced opioid consumption and therefore reduced opioid side effects. The investigators believe ultrasound guided TAP blocks will reduce pain and morphine consumption with a resultant improved patient satisfaction, earlier return of bowel function and earlier hospital discharge.

The key research question the investigators are trying to answer is whether TAP block provide better pain relief than local anaesthetic infiltration of the laparoscopic port sites. Both techniques are currently being used in our hospital and a retrospective audit demonstrated better analgesia and lower consumption of morphine in the TAP block group.The differences were not statistically significant as the number patients in the audit were not large enough.The investigators are hoping that this study will demonstrate that the difference is real by recruiting the necessary number of patients into each group (36 per group)

DETAILED DESCRIPTION:
Summary of Study Design The study will be a double blind randomised controlled trial with patients undergoing laparoscopic right hemicolectomy or laparoscopic high anterior resection randomly allocated into two groups, with the study group receiving bilateral TAP blocks followed by a morphine PCA and the control group receiving local anaesthetic infiltration of the laparoscopic port sites and specimen extraction site and a morphine PCA.

A double blind design was chosen to eliminate patient and observer bias in reporting of pain scores.

The presence of the control arm will ensure that any difference observed will be due to the effect of sensory nerve block due to the TAP block than due to the systemic effect of the injected local anaesthetic.

The null hypothesis will be that there is no difference between the groups in the amount of morphine consumed by the patients during 48 hours after the operation. We chose this measurement as an objective but indirect measurement of efficacy of TAP block and pain relief thus received. Measurement of pain with various scoring methods are reliable only when concurrent reduction in consumption of pain killers are demonstrated.

Recruitment and randomisation:

All patients meeting the inclusion criteria will receive a patient information leaflet and an invitation letter to participate in the study during the pre-assessment visit. We aim to recruit 72 patients (36 patients per group).

Informed consent will be taken by one of the investigators on the morning of the surgery, if the exclusion criteria are not applicable. Patients will be allotted consecutive participant numbers starting from one. Patients will be randomly allocated into either the study group and a control group. Randomisation will occur by using computer generated random numbers. Group allocation will be kept in a consecutively numbered, opaque, sealed envelope in the controlled drugs cupboard in theatre-6 anaesthetic room of Churchill hospital.Once patient has consented, the anaesthetist will open the corresponding numbered envelope and perform bilateral TAP blocks after induction of general anaesthesia, if the patient is in the study group the surgeons will infiltrate the port sites with local anaesthetic at the end of the procedure if the patient is in the control group.

Blinding:

The study group will receive bilateral TAP blocks with 20mls 0.25% bupivacaine on each side and the skin punctures on either sides will be covered with a small plaster. Patients in the control group will receive subcutaneous infiltration of the laparoscopic port sites and specimen extraction site with equivalent amount bupivacaine at the end of the procedure and small plasters will be stuck on either flanks approximately where the skin punctures for TAP block will be made.

The assessor of pain scores and morphine doses (Recovery nurse & Colo-rectal house officer) and the patient will be blinded to group allocation.

Patient: Plasters will be stuck on flanks of all the patients both study and control group so that patient will not know if they have received TAP block.

Recovery nurse: During handover to recovery the anaesthetist and scrub nurse will not mention about group allocation.

Colo-rectal house officer: The house officers( Junior Doctors) who will be following up in the ward will not present in the operating theatre, so they will be blinded

The study duration will be from induction of anaesthesia until the patients are medically fit for discharge from hospital. No extra visits other than routinely required for the surgical procedure is expected.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Undergoing elective laparoscopic high anterior resection without stoma or laparoscopic right hemicolectomy.
* American Society of Anaesthetists physical status (ASA) 1-3

Exclusion Criteria:

* Opioid tolerance
* Chronic abdominal pain
* Allergy/Intolerance: Morphine, local anaesthetics
* BMI>35 Kg/M2
* Previous major abdominal surgery
* High likelihood of conversion to open procedure
* Patients unable to communicate in written and spoken English
* Weight less than 50 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Crabtree, MB,ChB, FRCA, Principal Investigator — Nuffield Department of Anaesthetics, Oxford Radcliffe Hospitals NHS Trust , Oxford
Locations (1):
- The Churchill Hospital, Oxford Radcliffe Hospitals NHS trust, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Zafar N, Davies R, Greenslade GL, Dixon AR. The evolution of analgesia in an 'accelerated' recovery programme for resectional laparoscopic colorectal surgery with anastomosis. Colorectal Dis. 2010 Feb;12(2):119-24. doi: 10.1111/j.1463-1318.2009.01768.x. Epub 2009 Jan 16. PMID 19207712
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] McDonnell JG, O'Donnell BD, Farrell T, Gough N, Tuite D, Power C, Laffey JG. Transversus abdominis plane block: a cadaveric and radiological evaluation. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):399-404. doi: 10.1016/j.rapm.2007.03.011. PMID 17961838
- [Background] El-Dawlatly AA, Turkistani A, Kettner SC, Machata AM, Delvi MB, Thallaj A, Kapral S, Marhofer P. Ultrasound-guided transversus abdominis plane block: description of a new technique and comparison with conventional systemic analgesia during laparoscopic cholecystectomy. Br J Anaesth. 2009 Jun;102(6):763-7. doi: 10.1093/bja/aep067. Epub 2009 Apr 17. PMID 19376789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Started | 36 | 36
Completed | 28 | 28
Not Completed | 8 | 8
Not completed — Lost to Follow-up | 8 | 8

BASELINE CHARACTERISTICS:
Population: 8 cases converted to open and therefore excluded from analysis. 7 cases had incomplete and missing follow up data from the ward and were excluded from analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAP Block | Local Anaesthetic Infiltration | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 68.7 [65 to 75.5] | 67.8 [64.3 to 71.4] | 68.3 [64.3 to 75.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 16 | 13 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 28 | 28 | 56
BMI [Mean (Inter-Quartile Range); unit: Kg/m2] | 26.9 [22.4 to 27.3] | 28.9 [24.4 to 29.3] | 27.7 [22.9 to 29.1]

OUTCOME MEASURES:

1. Primary Outcome: Morphine Consumption in the First 48hours After the Operation
Description: Total morphine consumption in the first 48 hours after the surgery will be calculated from the drug chart and the Patient controlled analgesia(PCA)pump.
Time Frame: 48 hours after the operation
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 28 | 28
mg | 47.3 [36.2 to 58.5] | 46.7 [36.2 to 57.3]

2. Secondary Outcome: Numerical Rating Pain Scores at 48 Hours Postoperatively
Description: Numerical Rating Scores for Pain (0-10) 0= no pain 10= severe pain
Time Frame: 48 hours after the operation
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 28 | 28
units on a scale | 2 [1.5 to 5] | 2 [1 to 5]

3. Secondary Outcome: Nausea Score at 48 Hours Postoperatively
Description: 0-10 0= no nausea 10=severe nausea
Time Frame: 48 hours after the operation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 28 | 28
units on a scale | 0 [0 to 0] | 0 [0 to 0.25]

4. Secondary Outcome: Time to First Request for Rescue Analgesia
Description: The time will be calculated from the drug chart looking up when the first dose of rescue morphine was administered
Time Frame: After the operation patients will be followed up till they are medically fit to be discharged from the hospital an expected average of 5-7 days.
Population: data were not collected
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Mobilisation
Description: Time will be calculated from the nursing notes and patient diary, when the patient was first mobilised.
Time Frame: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 28 | 28
days | 1 [0.5 to 2] | 1 [0.5 to 2]

6. Secondary Outcome: Time to Successful Intake of Fluids
Description: Time will be calculated from the nursing notes and patient diary, when the patient had first successful intake of oral fluids.
Time Frame: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 28 | 28
days | 1.5 [0.5 to 3] | 2 [0.5 to 4]

7. Secondary Outcome: Time to Resumption of Normal Diet
Description: Time will be calculated from the nursing notes and patient diary, when the patient resumed normal diet.
Time Frame: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 28 | 28
days | 2 [1 to 5] | 2.5 [1 to 6]

8. Secondary Outcome: Time to First Bowel Motion
Description: Time will be calculated from the nursing notes and patient diary, when the patient had the first bowel motion.
Time Frame: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 28 | 28
days | 2.5 [1 to 5] | 3 [1 to 6]

9. Secondary Outcome: Time to First Flatus
Description: Time will be calculated from the nursing notes and patient diary, when the patient first passed flatus.
Time Frame: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 28 | 28
days | 1 [0.5 to 3] | 1 [0.3 to 3]

10. Secondary Outcome: Time to Medically Fit to Discharge
Description: Time will be calculated from the medical notes, when the decision that the patient is medically fit to be discharged was made.
Time Frame: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 28 | 28
days | 4.5 [3 to 9] | 4.5 [3 to 8]

11. Secondary Outcome: Total Morphine Consumption at 24hours
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: mg
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 28 | 28
mg | 30.9 [24 to 37.8] | 31 [24.1 to 37.9]

12. Secondary Outcome: Nausea at 24hours Post Operatively
Time Frame: 24 hours
Population: data lost during follow up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 21 | 23
units on a scale | 0 [0 to 0.5] | 0 [0 to 0]

13. Secondary Outcome: Time to Mobilization
Time Frame: days
Population: data lost in follow up
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 26 | 28
days | 1 [0.5 to 2] | 1 [0.5 to 2]

14. Secondary Outcome: Time to Hospital Discharge
Time Frame: days
Population: data lost on follow up
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Number analyzed (Participants) | 24 | 28
days | 4.5 [3 to 9] | 4.5 [3 to 8]

ADVERSE EVENTS:
Arm/Group | TAP Block | Local Anaesthetic Infiltration
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 0/36 | 0/35

LIMITATIONS AND CAVEATS:
Smaller number of subjects analysed than planned. Presented data should be carefully interpreted (and no conclusions should be drawn) since not enough patients were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes